CLINICAL TRIAL: NCT04223479
Title: Effect of Probiotic Supplementation on the Immune System in Patients With Ulcerative Colitis in Amman, Jordan
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Jordan (Other)
Responsible Party: Principal Investigator, Lana M. Agraib, Principal Investigator, University of Jordan
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2019/385
Record Dates: First submitted 2020-01-06; First posted 2020-01-10 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Ulcerative Colitis
Keywords: Ulcerative Colitis; immune system; Inflammatory markers; Probiotics
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Probiotic Formula Capsule (Experimental): In this intervention arm, the patients will receive oral viable capsules of probiotic contain (1*10 10 colony-forming unit (CFU)/g) of lactobacillus (Lactobacillus rhamnosus , Lactobacillus acidophilus, Lactobacillus reuteri, Lactobacillus paracasei, Lactobacillus casei, Lactobacillus gasseri, Lactobacillus plantarum) and bifidobacteria (Bifidobacterium lactis, Bifidobacterium breve, Bifidobacterium bifidum, Bifidobacterium longum, Bifidobacterium infantis) species three times a per day
  Interventions: Drug: Probiotic Formula Capsule
- Placebos (Placebo Comparator): In this intervention arm Placebo arm received three oral viable capsules daily, containing polysaccharides, without any viable probiotics matching the probiotic capsules in appearance, smell, and taste.
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Probiotic Formula Capsule — The Probiotic will be coded in a specific label by a researcher who will not be in contact with the participants and administrated randomly based on gender in a double-blind manner. The patient will receive 2 bottles of the drug every 2 weeks and will be followed weekly for 6 weeks.
  Other Names: Probiotics capsule; Probiotics supplement
  Arms: Probiotic Formula Capsule
Drug: Placebos — The Placebos will be coded in a specific label by a researcher who will not be in contact with the participants and administrated randomly based on gender in a double-blind manner. The patient will receive 2 bottles of the placebo every 2 weeks and will be followed weekly for 6 weeks.
  Other Names: Placebo oral capsule
  Arms: Placebos

SUMMARY:
Ulcerative colitis (UC) is a chronic Inflammatory bowel disease (IBD) that most likely results from the interaction between various environmental and genetic factors. Using probiotics as an adjunct to medical therapy might be useful in the treatment of UC and improving the symptoms of the disease. The result of studies that investigate the role of Probiotics supplementation in improving the inflammatory response, immune response and life quality of patients with the UC is not conclusive. So, this study aimed to study the effect of probiotics on the response of inflammatory markers, immune response, and quality of life in patients with UC.

An interventional double-blind randomized clinical trial (RCT) design will be used in this study. Forty patients will be recruited and randomly assigned to the placebo group (n=20) to receive 3 times a day placebo capsules; and probiotics group (n=20), to receive 3 times a day probiotic supplement. The demographic data, anthropometric measurements, IBD Quality of Life Questionnaire and blood samples will be collected at baseline and after 6 weeks of follow up. Interleukin-6, interleukin-1,interleukin-10 IL-10, C-reactive protein, tumor necrosis factor-alpha and complete blood count (CBC) will be measured.

The results will approve or disapprove the beneficial effect of using probiotics as adjuvant therapy for UC patients to raise the immune system as well as improving their quality of life.

DETAILED DESCRIPTION:
To meet the objectives of the study, an interventional double-blind randomized clinical trial (RCT) design will be used in this study. A placebo group will be included in parallel with the treatment group in this trail. Forty patients (aged 35-65 years) who diagnosed with mild to moderately active UC will be recruited conveniently from the gastroenterology section, the IBD clinic at the Jordan University Hospital, Amman, Jordan. Patients who meet the inclusion criteria and agree to participate will be centrally randomized to probiotic supplementation group or placebo group using computer-generated random numbers, that balanced allocation to groups A and B: in successive blocks each containing 20 patients each stratified by gender. The duration of the intervention will be 6 weeks.

For the participants, the Jordan University Hospital setting will be utilized for data collection. The patients will be recruited over 12 months and all patients will be asked to sign a written informed consent before enrollment. The patients will randomly be assigned to the placebo group (n=20), to receive 3 times a day placebo capsules contain polysaccharides, without any viable probiotics matching the probiotic capsules in appearance, smell, and taste; and probiotics group (n=20), to receive 3 times a day probiotic supplement. The administration of supplements will be under the supervision of the treating physician. The blood sample will be collected at baseline and at the end of 6 weeks of follow up.

The demographic data of each subject will be collected such as; gender, age, body mass index (BMI), tumor location, malignant tumors stage, tumor differentiation, educational level, occupation, family history, smoking, dietary and physical activity. At baseline and end of the follow-up, IBD Quality of Life Questionnaire will be collected and blood sample tests will be withdrawn and the following biochemical variables will be measured: immunoglobulin G, immunoglobulin M, immunoglobulin A, interleukin-6 (IL-6), C-reactive protein (CRP), interleukin-1(IL-1), interleukin-10(IL-10), interleukin-12 (IL-12), Tumor necrosis factor-alpha (TNF-α) and complete blood count (CBC).

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients,
* Age between 35 -65 years,
* Diagnosed with UC established by colonoscopy and histology, and suffering from mild to moderate UC as defined by Modified Mayo Disease Activity Index (MMDAI) (score 3-9).

Exclusion Criteria:

* Patients with age <35 years, >65 years,
* Pregnancy, planned pregnancy, breastfeeding women,
* Evidence of severe disease (MMDAI >10),
* Concurrent enteric infection,
* Use of antibiotics,
* Change in the dose of oral 5-aminosalicylic acid (5-ASA) within the past 4weeks, and use of rectal 5-ASA or steroids within 7 days before entry into the study,
* Received any investigational medicines within 3months,
* If they have significant hepatic, renal, endocrine, respiratory, neurological, or cardiovascular diseases

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-01-15 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-03-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed Isam Yamani, Pro.Dr, Study Chair — University of Jordan; Reema F Tayyem, Pro.Dr, Study Chair — University of Jordan
Locations (1):
- Jordan University Hospital, Amman, Jordan

IPD SHARING:
Plan to Share IPD: No
The center (Jordan University hospital) where the study conducted emphasis of maintaining privacy and confidentiality of the participants' data

REFERENCES:
- [Background] Abraham BP, Quigley EMM. Probiotics in Inflammatory Bowel Disease. Gastroenterol Clin North Am. 2017 Dec;46(4):769-782. doi: 10.1016/j.gtc.2017.08.003. Epub 2017 Oct 3. PMID 29173520
- [Background] Araya M, Morelli L, Reid G, et al. (2002), Guidelines for the evaluation of probiotics in food. Joint FAO/WHO Working Group report on drafting guidelines for the evaluation of probiotics in food, London; (ON, Canada). ftp://ftp.fao.org/es/esn/food/wgreport2.pdf (Accessed 19March, 2018).
- [Background] Bamias G, Corridoni D, Pizarro TT, Cominelli F. New insights into the dichotomous role of innate cytokines in gut homeostasis and inflammation. Cytokine. 2012 Sep;59(3):451-9. doi: 10.1016/j.cyto.2012.06.014. Epub 2012 Jul 12. PMID 22795953
- [Background] Bengtsson J, Adlerberth I, Ostblom A, Saksena P, Oresland T, Borjesson L. Effect of probiotics (Lactobacillus plantarum 299 plus Bifidobacterium Cure21) in patients with poor ileal pouch function: a randomised controlled trial. Scand J Gastroenterol. 2016 Sep;51(9):1087-92. doi: 10.3109/00365521.2016.1161067. Epub 2016 May 6. PMID 27150635
- [Background] Cai S, Kandasamy M, Rahmat JN, Tham SM, Bay BH, Lee YK, Mahendran R. Lactobacillus rhamnosus GG Activation of Dendritic Cells and Neutrophils Depends on the Dose and Time of Exposure. J Immunol Res. 2016;2016:7402760. doi: 10.1155/2016/7402760. Epub 2016 Jul 20. PMID 27525288
- [Background] Dargahi N, Johnson J, Donkor O, Vasiljevic T, Apostolopoulos V. Immunomodulatory effects of probiotics: Can they be used to treat allergies and autoimmune diseases? Maturitas. 2019 Jan;119:25-38. doi: 10.1016/j.maturitas.2018.11.002. Epub 2018 Nov 12. PMID 30502748
- [Background] de Moreno de Leblanc A, Del Carmen S, Zurita-Turk M, Santos Rocha C, van de Guchte M, Azevedo V, Miyoshi A, Leblanc JG. Importance of IL-10 modulation by probiotic microorganisms in gastrointestinal inflammatory diseases. ISRN Gastroenterol. 2011;2011:892971. doi: 10.5402/2011/892971. Epub 2011 Feb 8. PMID 21991534
- [Background] Feuerstein JD, Moss AC, Farraye FA. Ulcerative Colitis. Mayo Clin Proc. 2019 Jul;94(7):1357-1373. doi: 10.1016/j.mayocp.2019.01.018. PMID 31272578
- [Background] Gajendran M, Loganathan P, Jimenez G, Catinella AP, Ng N, Umapathy C, Ziade N, Hashash JG. A comprehensive review and update on ulcerative colitis. Dis Mon. 2019 Dec;65(12):100851. doi: 10.1016/j.disamonth.2019.02.004. Epub 2019 Mar 2. PMID 30837080
- [Background] Guandalini S, Sansotta N. Probiotics in the Treatment of Inflammatory Bowel Disease. Adv Exp Med Biol. 2019;1125:101-107. doi: 10.1007/5584_2018_319. PMID 30632114
- [Background] Kabeerdoss J, Devi RS, Mary RR, Prabhavathi D, Vidya R, Mechenro J, Mahendri NV, Pugazhendhi S, Ramakrishna BS. Effect of yoghurt containing Bifidobacterium lactis Bb12(R) on faecal excretion of secretory immunoglobulin A and human beta-defensin 2 in healthy adult volunteers. Nutr J. 2011 Dec 23;10:138. doi: 10.1186/1475-2891-10-138. PMID 22196482
- [Background] Kaplan GG, Ng SC. Globalisation of inflammatory bowel disease: perspectives from the evolution of inflammatory bowel disease in the UK and China. Lancet Gastroenterol Hepatol. 2016 Dec;1(4):307-316. doi: 10.1016/S2468-1253(16)30077-2. Epub 2016 Nov 10. PMID 28404201
- [Background] Konishi H, Fujiya M, Tanaka H, Ueno N, Moriichi K, Sasajima J, Ikuta K, Akutsu H, Tanabe H, Kohgo Y. Probiotic-derived ferrichrome inhibits colon cancer progression via JNK-mediated apoptosis. Nat Commun. 2016 Aug 10;7:12365. doi: 10.1038/ncomms12365. PMID 27507542
- [Derived] Rayyan YM, Agraib LM, Alkhatib B, Yamani MI, Abu-Sneineh AT, Tayyem RF. Does probiotic supplementation improve quality of life in mild-to-moderately active ulcerative colitis patients in Jordan? A secondary outcome of the randomized, double-blind, placebo-controlled study. Eur J Nutr. 2023 Oct;62(7):3069-3077. doi: 10.1007/s00394-023-03207-8. Epub 2023 Jul 27. PMID 37498369
- [Derived] Agraib LM, Yamani MI, Tayyem R, Abu-Sneineh AT, Rayyan YM. Probiotic supplementation induces remission and changes in the immunoglobulins and inflammatory response in active ulcerative colitis patients: A pilot, randomized, double-blind, placebo-controlled study. Clin Nutr ESPEN. 2022 Oct;51:83-91. doi: 10.1016/j.clnesp.2022.08.020. Epub 2022 Aug 20. PMID 36184252

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Assessed for eligibility (n=300)
  Excluded (n= 270)
  * Not meeting inclusion criteria (n=229)
  * Declined to participate (n=15)
  * Other reasons (n=26)
  Randomized (n=30)
Groups:
- Placebo Group: In this intervention arm Placebo arm received three oral viable capsules daily, containing polysaccharides, without any viable probiotics matching the probiotic capsules in appearance, smell, and taste.
  Placebos: The Placebos will be coded in a specific label by a researcher who will not be in contact with the participants and administrated randomly based on gender in a double-blind manner. The patient will receive 2 bottles of the placebo every 2 weeks and will be followed weekly for 6 weeks.
- Probiotic Group: In this intervention arm, the patients will receive oral viable capsules of probiotic contain (1*10 10 colony-forming unit (CFU)/g) of lactobacillus (Lactobacillus rhamnosus , Lactobacillus acidophilus, Lactobacillus reuteri, Lactobacillus paracasei, Lactobacillus casei, Lactobacillus gasseri, Lactobacillus plantarum) and bifidobacteria (Bifidobacterium lactis, Bifidobacterium breve, Bifidobacterium bifidum, Bifidobacterium longum, Bifidobacterium infantis) species three times a per day
  Probiotic Formula Capsule: The Probiotic will be coded in a specific label by a researcher who will not be in contact with the participants and administrated randomly based on gender in a double-blind manner. The patient will receive 2 bottles of the drug every 2 weeks and will be followed weekly for 6 weeks.
Period: Overall Study
Arm/Group | Placebo Group | Probiotic Group
Started | 16 | 14
Completed | 12 | 12
Not Completed | 4 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Probiotic Formula Capsule | Placebos | Total
Number analyzed (Participants) | 16 | 14 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 16 | 14 | 30
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 8 | 18
  Male | 6 | 6 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 16 | 14 | 30
Region of Enrollment [Number; unit: participants]
  Jordan | 16 | 14 | 30
Ethnicity [Count of Participants; unit: Participants]
  Arabs | 16 | 14 | 30
  Others | 0 | 0 | 0
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 25.3 (6.8) | 24.6 (5.7) | 24.95 (6.25)
Family history of IBD [Count of Participants; unit: Participants]
  Yes | 5 | 2 | 7
  No | 11 | 12 | 23
History of Probiotic use [Count of Participants; unit: Participants]
  Yes | 1 | 2 | 3
  No | 15 | 12 | 27

OUTCOME MEASURES:

1. Primary Outcome: The Level of Immunoglobulin (Ig) A
Description: The level of Immunoglobulin (Ig) A in mg/dL was tested at the end of follow-up (after 6 weeks of follow-up) based on an Immunoturbidimetric assay using Cobas-C501
Time Frame: at the end of 6 weeks of follow-up
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo Group | Probiotic Group
Number analyzed (Participants) | 12 | 12
mg/dL | 270.42 (71.79) | 208.63 (85.84)

2. Primary Outcome: The Level of Immunoglobulin (Ig) G
Description: The level of Immunoglobulin (Ig) G in mg/dL was tested at the end of follow-up (after 6 weeks of follow-up) based on an Immunoturbidimetric assay using Cobas-C501
Time Frame: at the end of 6 weeks of follow up
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo Group | Probiotic Group
Number analyzed (Participants) | 12 | 12
mg/dL | 1267.36 (177.6) | 1214.70 (236.3)

3. Primary Outcome: The Level of Immunoglobulin (Ig) M
Description: The level of Immunoglobulin (Ig) M in mg/dL was tested at the end of follow-up (after 6 weeks of follow-up) based on an Immunoturbidimetric assay using Cobas-C501
Time Frame: at the end of 6 weeks of follow-up
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo Group | Probiotic Group
Number analyzed (Participants) | 12 | 12
mg/dL | 114.64 (62.03) | 104.10 (39.57)

4. Primary Outcome: The Level of Interleukin (IL)-6
Description: The Level of Interleukin (IL)-6 in pg/ml measured aat the end of follow-up (after 6 weeks of follow-up) by a two-site sandwich Enzyme-Linked Immunosorbent Assay (ELISA)
Time Frame: at the end of 6 weeks of follow-up
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Placebo Group | Probiotic Group
Number analyzed (Participants) | 12 | 12
pg/ml | 10.84 (3.30) | 9.40 (3.13)

5. Primary Outcome: The Level of Interleukin (IL)-1
Description: The Level of Interleukin (IL)-1 in pg/ml measured at the end of follow-up (after 6 weeks of follow-up) by a two-site sandwich Enzyme-Linked Immunosorbent Assay (ELISA)
Time Frame: at the end of 6 weeks of follow-up
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Placebo Group | Probiotic Group
Number analyzed (Participants) | 12 | 12
pg/ml | 7.33 (3.31) | 8.55 (3.45)

6. Primary Outcome: The Level of Interleukin (IL)-10
Description: The Level of Interleukin (IL)-10 in pg/ml was measured at the end of follow-up (after 6 weeks of follow-up) by a two-site sandwich Enzyme-Linked Immunosorbent Assay (ELISA)
Time Frame: at the endo f 6 weeks of follow-up
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Placebo Group | Probiotic Group
Number analyzed (Participants) | 12 | 12
pg/ml | 22.89 (12.49) | 37.10 (14.95)

7. Primary Outcome: The Level of Tumor Necrosis Factor (TNF)-α
Description: The Level of TNF-α in pg/ml measured at the end of follow-up (after 6 weeks of follow-up) by a two-site sandwich Enzyme-Linked Immunosorbent Assay (ELISA)
Time Frame: at the endo of 6weeks of follow-up
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Placebo Group | Probiotic Group
Number analyzed (Participants) | 12 | 12
pg/ml | 9.36 (1.57) | 9.58 (1.75)

8. Primary Outcome: The Level of C-reactive Protein (CRP)
Description: The Level of CRP in mg/ml measured at the end of follow-up (after 6 weeks of follow-up) based on an Immunoturbidimetric assay using Cobas-C501
Time Frame: at the end of 6 weeks of follow-up
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Placebo Group | Probiotic Group
Number analyzed (Participants) | 12 | 12
mg/L | 4.65 (0.24) | 4.54 (0.14)

9. Secondary Outcome: Quality of Life of Patients
Description: The average score of the general quality of life (QoL) subscales was assessed by the Short Quality of Life in Inflammatory Bowel Disease Questionnaire (SIBDQ). The SIBDQ contains 10 questions for 4 functional scales (Bowel, Systemic, emotional, and social). For each question, there a regraded responses on a 7-point Likert scale ranging from one (representing the ''worst'' aspect) to seven (representing the ''best'' aspect). Total SIBDQ scores range from 10 to 70.Higher scores reflect better well-being.
Time Frame: at the end of 6 weeks of follow-up
Measure: Mean (Standard Deviation); unit: points
Arm/Group | Placebo Group | Probiotic Group
Number analyzed (Participants) | 12 | 12
points | 4.96 (1.27) | 6.54 (0.29)

10. Other Pre Specified Outcome: The Level of White Blood Cell Count (WBC)
Description: The level of WBC as cells*10^9/l measured at the end of follow-up (after 6 weeks of follow-up) using the automated analyzer Sysmex XS-500i
Time Frame: at the end of 6 weeks of follow-up
Measure: Mean (Standard Deviation); unit: cells10^9/l
Arm/Group | Placebo Group | Probiotic Group
Number analyzed (Participants) | 12 | 12
cells10^9/l | 8.18 (2.90) | 6.72 (2.01)

11. Other Pre Specified Outcome: The Level of Red Blood Cell Count (RBC)
Description: The level of RBC as cells*10^12/l measured at the end of follow-up (after 6 weeks of follow-up) using the automated analyzer Sysmex XS-500i
Time Frame: at the end of 6 weeks of follow-up
Measure: Mean (Standard Deviation); unit: cells10^12/ul
Arm/Group | Placebo Group | Probiotic Group
Number analyzed (Participants) | 12 | 12
cells10^12/ul | 4.73 (0.55) | 4.95 (0.36)

12. Other Pre Specified Outcome: The Mean Corpuscular Volume (MCV)
Description: The MCV in fl measured at the end of follow-up (after 6 weeks of follow-up) using the automated analyzer Sysmex XS-500i
Time Frame: at the end of 6 weeks of follow-up
Measure: Mean (Standard Deviation); unit: fl
Arm/Group | Placebo Group | Probiotic Group
Number analyzed (Participants) | 12 | 12
fl | 85.68 (9.23) | 83.63 (7.33)

13. Other Pre Specified Outcome: The Mean Corpuscular Hemoglobin (MCH)
Description: The MCH in pg measured at the end of follow-up (after 6 weeks of follow-up) using the automated analyzer Sysmex XS-500i
Time Frame: at the end of 6 weeks of follow-up
Measure: Mean (Standard Deviation); unit: pg
Arm/Group | Placebo Group | Probiotic Group
Number analyzed (Participants) | 12 | 12
pg | 28.70 (3.27) | 27.88 (2.96)

14. Other Pre Specified Outcome: The Mean Corpuscular Hemoglobin Concentration (MCHC)
Description: The MCH in g/dl measured at the end of follow-up (after 6 weeks of follow-up) using the automated analyzer Sysmex XS-500i
Time Frame: at the end of 6 weeks of follow-up
Measure: Mean (Standard Deviation); unit: g/dl
Arm/Group | Placebo Group | Probiotic Group
Number analyzed (Participants) | 12 | 12
g/dl | 33.28 (0.90) | 33.52 (1.31)

15. Other Pre Specified Outcome: The Platelet Count
Description: The Platelet count as cells 10^9/ll measured at the end of follow-up (after 6 weeks of follow-up) using the automated analyzer Sysmex XS-500i
Time Frame: at the end of 6 weeks of follow-up
Measure: Mean (Standard Deviation); unit: cells*10^9/l
Arm/Group | Placebo Group | Probiotic Group
Number analyzed (Participants) | 12 | 12
cells*10^9/l | 292.40 (72.05) | 288.18 (69.47)

16. Other Pre Specified Outcome: The of Hemoglobin
Description: The Hemoglobin in g/dl measured at the end of follow-up (after 6 weeks of follow-up) using the automated analyzer Sysmex XS-500i
Time Frame: at the end of 6 weeks of follow-up
Measure: Mean (Standard Deviation); unit: g/l
Arm/Group | Placebo Group | Probiotic Group
Number analyzed (Participants) | 12 | 12
g/l | 13.54 (2.01) | 13.78 (1.54)

17. Other Pre Specified Outcome: The Mean Platelet Volume (MPV)
Description: The MPV in fl measured at the end of follow-up (after 6 weeks of follow-up) using the automated analyzer Sysmex XS-500i
Time Frame: at the end of 6 weeks of follow-up
Measure: Mean (Standard Deviation); unit: fl
Arm/Group | Placebo Group | Probiotic Group
Number analyzed (Participants) | 12 | 12
fl | 10.67 (1.22) | 10.71 (0.83)

18. Other Pre Specified Outcome: The Level of Lymphocytes
Description: The number of lymphocytes cells as cells*10^9/L measuredat the end of follow-up (after 6 weeks of follow-up) using the automated analyzer Sysmex XS-500i
Time Frame: at the end of 6 weeks of follow-up
Measure: Mean (Standard Deviation); unit: cells*10^9/L
Arm/Group | Placebo Group | Probiotic Group
Number analyzed (Participants) | 12 | 12
cells*10^9/L | 2.50 (0.93) | 2.40 (0.69)

19. Other Pre Specified Outcome: The Level of Monocytes
Description: The number of Monocytes cells measured at the end of follow-up (after 6 weeks of follow-up) using the automated analyzer Sysmex XS-500i
Time Frame: at the end of 6 weeks of follow-up
Measure: Mean (Standard Deviation); unit: cells10^9/l
Arm/Group | Placebo Group | Probiotic Group
Number analyzed (Participants) | 12 | 12
cells10^9/l | 0.67 (0.28) | 0.59 (0.16)

20. Other Pre Specified Outcome: The Level of Eosinophils
Description: The number of eosinophils cells measured at the end of follow-up (after 6 weeks of follow-up) using the automated analyzer Sysmex XS-500i
Time Frame: at the end of 6 weeks of follow-up
Measure: Mean (Standard Deviation); unit: cells10^9/l
Arm/Group | Placebo Group | Probiotic Group
Number analyzed (Participants) | 12 | 12
cells10^9/l | 0.25 (0.19) | 0.15 (0.10)

21. Other Pre Specified Outcome: The Level of Basophils
Description: The number of basophils cells measured at the end of follow-up (after 6 weeks of follow-up) using the automated analyzer Sysmex XS-500i
Time Frame: at the end of 6 weeks of follow-up
Measure: Mean (Standard Deviation); unit: cells10^9/l
Arm/Group | Placebo Group | Probiotic Group
Number analyzed (Participants) | 12 | 12
cells10^9/l | 0 (0) | 0 (0)

22. Other Pre Specified Outcome: The Level of Neutrophils
Description: The number of neutrophils cells measured at the end of follow-up (after 6 weeks of follow-up) using the automated analyzer Sysmex XS-500i
Time Frame: at the end of 6 weeks of follow-up
Measure: Mean (Standard Deviation); unit: cells10^9/l
Arm/Group | Placebo Group | Probiotic Group
Number analyzed (Participants) | 12 | 12
cells10^9/l | 5.05 (2.35) | 3.56 (1.59)

ADVERSE EVENTS:
Time Frame: two month period for each patient
Description: Non
Arm/Group | Probiotic Formula Capsule | Placebos
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-09-22): https://cdn.clinicaltrials.gov/large-docs/79/NCT04223479/Prot_000.pdf
  • Statistical Analysis Plan (2023-11-22): https://cdn.clinicaltrials.gov/large-docs/79/NCT04223479/SAP_001.pdf